CLINICAL TRIAL: NCT05791669
Title: Arrest of Interproximal Caries Lesion in Primary Molars With 38% Silver Diamine Fluoride Solution and 5% Sodium Fluoride Varnish: A Randomized Clinical Trial
Brief Title: Arrest of Interproximal Caries Lesion With 38% Silver Diamine Fluoride Solution
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PGIDS/BHRC/21/13
Record Dates: First submitted 2022-11-12; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2022-11

CONDITIONS: Caries Arrested
Keywords: Caries arrest ,interproximal caries, primary molars, SDF
MeSH Terms: interventions — silver diamine fluoride; Bifluorid 12

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 38% silver diamine fluoride (Experimental)
  Interventions: Drug: Silver diamine fluoride
- 5% sodium fluoride varnish (Active Comparator)
  Interventions: Drug: Sodium fluoride varnish

INTERVENTIONS:
Drug: Silver diamine fluoride — Silver diamine fluoride is a topical medication composed of 25% silver, 5% fluoride, 8% ammonia, and 62% Deionized water, used to treat and prevent dental caries and relieve dentinal hypersensitivity.
  Other Names: FAgamin SDF38%
  Arms: 38% silver diamine fluoride
Drug: Sodium fluoride varnish — It is a topical application with an active ingredient of 5% sodium fluoride(22,600ppm fluoride).it prolongs the contact time between the fluoride and tooth surface and promotes remineralization and inhibits demineralization.
  Other Names: VOCO profluorid varnish
  Arms: 5% sodium fluoride varnish

SUMMARY:
This study was conducted to assess the efficacy of 38% Silver Diamine fluoride and compare it with 5% sodium fluoride varnish in arresting interproximal caries in primary molars at 12 months follow-up. Bitewing radiographs were taken to diagnose as well as to assess caries depth at follow up visits. Each bitewing was scored based on ICCMS radiographic criteria and was compared (follow-ups to baseline)to check for caries arrest.

Interproximal caries included in this study, according to ICCMS criteria, were at stages- RA - caries limited to outer half of enamel RA2 - caries limited to the inner half of enamel RA3 - caries limited to outer third of dentine RA4 - caries limited to middle third of dentine

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 5 to 9 years.
2. Presence of at least 2 primary molars with interproximal caries.
3. Carious lesions of enamel or outer or middle third of dentin in primary molars, as assessed by bitewing radiographs with ICCMSTM scoring (RA1, RA2, RA3, RB4).

Exclusion Criteria:

1. Presence of advanced carious lesions reaching inner third of dentin detected by bitewing radiographic examinations ICCMSTM (RC5, RC6).

3. Children or adolescents that refuse to participate in the study or present negative behaviours.

4. Teeth with premature hypermobility 5. Both physically and mentally disabled children

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Caries arrest | 12 months
  Assessment with bitewing radiographs based on ICCMS radiographic scoring system

CONTACTS AND LOCATIONS:
Locations (1):
- Post graduate institute of dental sciences, Rohtak, Haryana, India